CLINICAL TRIAL: NCT04067245
Title: The Use of Tetrasodium EDTA Catheter Lock Solution for Patients on Home Parenteral Nutrition: Ease of Use and Cost Analysis
Brief Title: Use of Tetrasodium EDTA Catheter Lock Solution for Patients on HTPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Johane Allard, Senior Researcher at University of Toronto, Gastroenterologist at University Health Network, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-6325.0
Record Dates: First submitted 2019-04-25; First posted 2019-08-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Catheter Complications
Keywords: Home Total Parenteral Nutrition; Tetrasodium EDTA catheter lock solution; Catheter Complications; Catheter-Related Thrombosis; Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tetrasodium EDTA cathether lock solution (Other): There is only one arm in this study where home parenteral nutrition patients who meet the inclusion criteria will receive tetrasodium EDTA catheter lock solution.
  Interventions: Device: Tetrasodium EDTA catheter lock solution

INTERVENTIONS:
Device: Tetrasodium EDTA catheter lock solution — Home parenteral nutrition patients who meets inclusion criteria is to receive tetrasodium edta catheter lock solution. Patient will receive standard catheter lock solution of heparin/saline for 1 month, followed by tetrasodium EDTA catheter lock solution using withdrawal method for 1 month and followed by tetrasodium EDTA catheter lock solution using flush method for 1 month. In total, patient will stay in the study for 3 months. A phone call will be conducted before the start of the study to give instruction to patient regarding the use of catheter lock solution. Time taken to connect and disconnect TPN will be recorded by patients, twice a month on first and last mondays of the month for 3 months. A survey regarding the ease of use of catheter lock solution will be conducted at the end of each month via phone by nurse coodinator.

SUMMARY:
Parenteral nutrition (PN) is a lifesaving therapy in patients with chronic intestinal failure. PN is administered via a central venous catheter (CVC), and patients are dependent on this line for ongoing nutrition. However, the presence of a CVC is associated with a risk of thrombosis and bloodstream infection. Many different types of catheter lock solutions have been used to mitigate these risks. They include solutions primarily aimed at reducing thrombosis, such as heparin and citrate, and others primarily aimed at reducing infection such as ethanol and antibiotics (for example, taurolidine). One recently developed solution, tetrasodium EDTA, aims to reduce both thrombosis and infection. This scientific review provides an overview of central venous catheter lock solutions, and an ease-of-use and cost analysis comparing heparin and tetrasodium EDTA in one home parenteral nutrition program in Toronto, Canada.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) is a life-sustaining therapy required in patients who do not have a functioning gastrointestinal tract. This can be either second to surgical removal, or malfunction (such as in malabsorptive conditions and dysmotility). The intravenous provision of nutrition requires central venous access where a hyperosmolar nutrient solution can be infused. A variety of central venous catheters (CVCs) can be used, including peripherally inserted central catheters (PICC), tunneled catheters and implanted ports. The most common complication, and most frequent cause of hospitalization in patients on home PN is bloodstream infection.

There are several new devices or solutions that are being developed to be used as primary prophylaxis for CRBSI. These include catheters with antibacterial and/or anti-biofilm properties and different catheter lock solutions. Antibiotic lock solutions have been used for salvage of central venous catheters in confirmed CRBSI. However, it is not recommended as a primary prophylaxis due to the creation of resistant organisms. According to the United States Center for Disease Control (CDC), antibiotics 'should be used only to manage infection.' However, one antimicrobial solution, taurolidine, has not been found to promote the emergence of resistant bacterial strains and it has been used successfully as a lock solution to prevent CRBSI. Although an antibiotic may have anti-biofilm properties in high concentrations but it does not have anticoagulant properties. Ethanol lock solutions (varying concentrations, but usually 70%) have also been used successfully to reduce CRBSI, however, there have been adverse events when they are used in polyurethane lines and it does not inherently have anticoagulant properties. Historically, citrate lock solution has also been used to maintain catheter patency, but in a meta-analysis, there was no difference between heparin and citrate lock with regards to catheter thrombosis or catheter related bloodstream infection.

Although its use has been evaluated in hemodialysis catheters, there are no known studies examining the use of a tetra-sodium EDTA catheter lock solution in central venous catheters of patients on home PN. Although both hemodialysis and home PN require central venous catheters, there are many differences inherent to the different usages. First, the types of catheters that are used can differ. There is more variety in the types of catheters used for home PN. Second, most patients undergo hemodialysis on a fixed schedule, three times per week for 4 to 8 hours each time, and, for the majority of patients, this is done in-center, with the assistance of a nurse. On the other hand, home PN is usually administered five or more days per week, at home, over 12 or more hours. It can be either administered with the assistance of a home care nurse or by the patient and/or their family/partner. Furthermore, the substance infused through the catheter is different. Specifically, amino acids and fat emulsions are usually only infused in home PN, although electrolytes and fluids can be infused in both.

Kitelock™, 4% tetrasodium EDTA catheter lock solution is the sole product of SterileCare Inc, a private medical devices and equipment company registered federally in Canada, and based in Markham, Ontario. Kitelock™ is licensed as a medical device, class 2 (license #96962, issue date 2016-05-10), by Health Canada.

The aim of this study is to perform cost- and ease-of-use analyses in patients on home parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Adult over the age of 18
* Both males and females
* Clinically stable for at least 4 weeks with no acute medical co-morbidities

Exclusion Criteria:

* Inability to give informed consent
* Alcohol or drug abuse
* Pregnant and lactating women
* Clinical instability such as the following:
* Acute pulmonary edema
* Decompensated heart failure
* Decompensated chronic liver disease
* Severe post-traumatic conditions
* Uncontrolled diabetes mellitus
* Acute myocardial infarction
* Acute stroke
* Acute thromboembolism
* Metabolic acidosis
* Sepsis
* Hypotonic dehydration
* Coagulopathy with prolonged aPTT or INR
* Unstable oncology patient
* Subjects who are hypersensitive or allergic to the product ingredients of tetrasodium EDTA
* Active therapy with long-term anti-microbial, such as taurolidine (not including patients receiving intermitted antimicrobial treatment for small intestinal bacterial overgrowth)
* Active participation in another home TPN clinical trial which may interfere with the results

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Ease of use | 24 months
  Acceptability of the new catheter lock solution by administering a questionnaire survey that will be conducted by the end of the usage. The questionnares will require the participant to rate the overall satisfaction of the product as '1. unsatisfied or 2. neutral or 3. satistified' and to rate the amount of time it takes to prepare the product as '1. took long or 2. neutral or 3. doesn't take too long and 3rd question compared to usual product (heparin), how easy is this product as '1. harder than heparin or 2. the same or 3. easier than heparin' and last question is ask if participant would continue to use this lock solution 'Yes' or 'No' and why not?

SECONDARY OUTCOMES:
Time taken to use the catheter lock | 24 months
  To evaluate time required to use the catheter lock solution by recording time taken to connect and disconnect TPN on the first and last Monday of every month.
Cost analysis | 24 months
  Cost analysis of using tetrasodium EDTA catheter lock solution versus heparin saline catheter lock solution

CONTACTS AND LOCATIONS:
Overall Officials: Ennaliza Salazar, Study Chair — TPN team
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Percival SL, Kite P, Eastwood K, Murga R, Carr J, Arduino MJ, Donlan RM. Tetrasodium EDTA as a novel central venous catheter lock solution against biofilm. Infect Control Hosp Epidemiol. 2005 Jun;26(6):515-9. doi: 10.1086/502577. PMID 16018425
- [Background] Kanaa M, Wright MJ, Akbani H, Laboi P, Bhandari S, Sandoe JA. Cathasept Line Lock and Microbial Colonization of Tunneled Hemodialysis Catheters: A Multicenter Randomized Controlled Trial. Am J Kidney Dis. 2015 Dec;66(6):1015-23. doi: 10.1053/j.ajkd.2015.04.047. Epub 2015 Jun 30. PMID 26141306
- [Background] Banfi G, Salvagno GL, Lippi G. The role of ethylenediamine tetraacetic acid (EDTA) as in vitro anticoagulant for diagnostic purposes. Clin Chem Lab Med. 2007;45(5):565-76. doi: 10.1515/CCLM.2007.110. PMID 17484616
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC). Guidelines for the prevention of intravascular catheter-related infections. Clin Infect Dis. 2011 May;52(9):e162-93. doi: 10.1093/cid/cir257. Epub 2011 Apr 1. No abstract available. PMID 21460264
- [Background] Zhao Y, Li Z, Zhang L, Yang J, Yang Y, Tang Y, Fu P. Citrate versus heparin lock for hemodialysis catheters: a systematic review and meta-analysis of randomized controlled trials. Am J Kidney Dis. 2014 Mar;63(3):479-90. doi: 10.1053/j.ajkd.2013.08.016. Epub 2013 Oct 11. PMID 24125729

DOCUMENTS (1):
  • Study Protocol (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT04067245/Prot_000.pdf